CLINICAL TRIAL: NCT07145190
Title: SL-APO in the Treatment of Patients With Parkinson's Disease: a Real-world Evidence Study to Identify Titration and Usage Schemes - SL-START
Brief Title: SL-START - SubLingual Apomorphine Schemes of TitrAtion in Real-world Treatment
Status: Recruiting | Type: Observational
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIA-KYNMB-401
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
Keywords: Kynmobi; SL-APO
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SL-START: SL-APO is available as a treatment initiation pack, containing two sublingual films of each strength (total of 30 films). The treatment initiation pack is usually used at the start of treatment to find an effective and tolerable dose. Depending on the patient response, not all doses in this pack may be needed.
  Interventions: Drug: SL-APO

INTERVENTIONS:
Drug: SL-APO — Patients should start with a dose of 10 mg SL-APO. Dose initiation should occur when the patient is having an OFF episode. If the patient tolerates the 10 mg dose, and responds adequately (meaning satisfactory motor response within 30 minutes), the maintenance dose should be 10 mg. If the dose is tolerated but the response is insufficient, continue to titrate in 5 mg increments when the patient is having an OFF episode and assess response until an effective and tolerable dose is achieved, up to a maximum of 30 mg per dose and up to five times a day. If an "ON" response is achieved and if clinically warranted, consider the need to further up-titrate as tolerated to achieve a better "ON" response. The minimal interval between doses is 2 hours, with no more than one dose of SL-APO per OFF episode.
  Other Names: Kynmobi

SUMMARY:
The purpose of the study is to generate real-world evidence data for the on-demand treatment with SL-APO, focusing on understanding its usage and titration practices including individual dose determination after dose-adjustment to ultimately understand their influence in patient satisfaction, treatment persistence, and the balance between effectiveness and safety. The data may help optimize titration approaches to better meet the patient's needs.

DETAILED DESCRIPTION:
This study is a prospective, observational, real-word evidence study. It is a non-interventional study according to article 2(4) of the Clinical Trials Regulation. Visits are documented as they occur in the routine of the practice or PD clinic.

The medical evaluation that leads to a treatment plan for the patient is not part of this study. The treatment plan may not include SL-APO. This study protocol becomes relevant only after unbiased prescription of SL-APO. Under no circumstances will access to treatment be contingent upon participation in the study. No additional procedures or examinations are required besides the ones already performed per local medical practice.

Patients who will initiate SL-APO according to the SmPC are potential study patients. After the patient's consent to participate in the study, the study starts with the baseline visit at the site (dark blue icon). The tolerance and efficacy of 10 mg SL-APO is tested for a patient in the OFF-state. In case of an insufficient "ON"-response of the first 10 mg dose, dose finding continues with titration at home (light blue house). The Titration follow-up (FU) takes place during the dose finding phase preferably when the patient has reached the preferred dose. The Titration FU can take place as a call or on-site. If a patient is not in the optimal dose during the Titration FU, they will be called again, as per their practice routine. Note, the only data collected from the Titration FU is if the optimal dose according to the HCP has been reached (and the date of the call). Patients will keep a Patient Titration Diary from the baseline visit to the end of titration. The diary entries are started from the 2nd intake of SL-APO. This is regardless of whether the intake takes place at home or in the clinical environment. Patients will keep a Patient Maintenance Diary after the end of titration until the end of the study. For at least the first 7 days and a minimum of 10 intakes, the Patient Maintenance Diary is kept daily, followed by a weekly entry. At 3 and 6 months, FU visits take place at the site. The 6-month FU visit marks the end of the study. The Investigator will decide if patients should continue to be prescribed the maintenance dose after the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years of age.
* The patient has a clinical diagnosis of idiopathic Parkinson's disease.
* The patient will initiate SL-APO for the treatment of OFF episodes according to the SmPC.
* The patient is not currently on titration or maintenance dose for SL-APO.
* The patient has provided written informed consent to participate in this study.

Exclusion Criteria:

* The patient is participating in a clinical trial with an investigational drug.
* The patient has presented with dementia or evidence of cognitive decline as determined by the investigator.
* The patient has a history of psychotic disorder.
* The patient presents any other contraindication according to the SL-APO SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients experiencing OFF symptoms which cannot be managed by oral anti-PD medication. For clarification, patients who have previously been exposed to apomorphine can also be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Identify the most frequent dose used after dose-adjustment | Up to 6 months
  The purpose of the study is to generate real-world evidence data for the on-demand treatment with SLAPO, focusing on understanding its usage and titration practices including individual dose determination after dose-adjustment to ultimately understand their influence in patient satisfaction, treatment persistence, and the balance between effectiveness and safety. The data may help optimize titration approaches to better meet the patient's needs.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kassubek, Prof Dr med, Principal Investigator — Praxis für Neurologie und Geriatrie (Ulm)
Locations (12):
- Germany (12):
  - Charité - Universitätsmedizin Berlin - Sektion für Bewegungsstörungen und Neuromodulation, Berlin
  - Alexianer St. Joseph Berlin-Weißensee GmbH, Berlin
  - Praxis für Neurologie, Berlin
  - Katholisches Klinikum Bochum gGmbH, Universitätsklinikum St.Josef-Hospital, Klinik für Neurologie, Bochum
  - UNIVERSITÄTSKLINIKUM FREIBURG - Neurozentrum Klinik für Neurologie und Neurophysiologie im Neurozentrum, Freiburg im Breisgau
  - Praxis für Neurologie und Psychiatrie, Fulda
  - Klinik am Tharandter Wald, Hetzdorf
  - Klinik für Neurologie und Neurologische Frührehabilitation, Osnabrück
  - Die Nerven Docs, Siegen
  - Neurologische Klinik Sorpesee, Sundern
  - Praxis für Neurologie und Geriatrie, Ulm
  - Neurologie am Funkerberg, Wusterhausen

IPD SHARING:
Plan to Share IPD: No